CLINICAL TRIAL: NCT01085422
Title: A Pilot Study Combining ABT-888, an Oral PARP Inhibitor, With Temozolomide in Patients With Metastatic Castration Resistant Prostate Cancer Who Have Failed Up to Two Non-hormonal Systemic Therapies
Brief Title: A Study Combining ABT-888, Oral PARP Inhibitor, With Temozolomide in Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-070
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — veliparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: ABT-888; Drug: temozolomide

INTERVENTIONS:
Drug: ABT-888 — Subjects will be given ABT-888 on Days 1 -7 every 28 days orally and temozolomide on days 1-5 on days 1-5 every 28 days orally with ABT-888
  Other Names: ABT-888, veliparib
Drug: temozolomide — Subjects will be given ABT-888 40 mg twice daily on Days 1 -7 every 28 days orally and temozolomide on days 1-5 every 28 days orally with ABT-888

SUMMARY:
Assess whether the combination of ABT-888 with temozolomide (TMZ) has activity in subjects with metastatic castration resistant prostate cancer (CRPC) as reflected by the prostate-specific antigen (PSA) response.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically or cytologically confirmed prostate cancer.
* Metastatic prostate cancer with measurable and/or bony disease that has progressed despite androgen deprivation therapy and at least one and no more than two prior systemic non hormonal therapies (at least one must include docetaxel) for castration resistant metastatic disease.
* At least 28 days must have elapsed since completion of prior anti-cancer therapy and must have recovered from all side effects to < Grade 1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. ECOG PS 3 is allowed if due to pain.
* Subjects must have PSA progression defined as:

  * A 25% increase in PSA over a baseline value with an increase in the absolute value of PSA level by 2 ng/ml, that is confirmed by another PSA level at a minimum of 1 week interval.
* Subjects must have a minimum PSA of > 2 ng/ml.
* Testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with a luteinizing hormone-releasing hormone (LHRH) analogue if they have not undergone orchiectomy.
* No investigational or commercial agents (other than LHRH analogue) or therapies including other hormonal agents such as antiandrogens or herbal medications may be administered with the intent to treat the subject's malignancy. Subjects on stable doses of steroids or megestrol acetate (for hot flashes or appetite) are allowed.
* Four weeks must have elapsed since major surgery.
* Prior radiotherapy is allowed as long as the bone marrow function is adequate and at least 4 weeks has elapsed since completion of radiation therapy. No prior radiopharmaceuticals are allowed.
* Subjects must have normal organ and bone marrow function as defined below obtained within two weeks from treatment initiation:

  * Bone Marrow: absolute neutrophil count ≥ 1,500/mcL; platelets ≥ 100,000/mcL; hemoglobin ≥ 9.0 g/dL
  * Renal function: Serum creatinine ≤ 1.5 × upper limits of institution's normal (ULIN) range or creatinine clearance ≥ 50 mL/min/1.73 m2
  * Hepatic Function: Aspartate aminotransferase (AST) and/or alanine transaminase (ALT) ≤ 2.5 × ULIN. For subjects with liver metastases, AST and/or ALT < 5 × ULIN. Bilirubin ≤ 1.5 × ULIN (Subjects with Gilbert's Syndrome may have a bilirubin ≥ 1.5 × ULIN)
* Subjects who refuse to provide blood samples for the correlative studies will be eligible.
* ABT-888 and temozolomide are known to be teratogenic, therefore men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Subjects with treated and controlled epidural disease are permitted into the study.
* Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.

Exclusion Criteria:

* A subject with cord compression or a history of uncontrolled central nervous system (CNS) metastases or leptomeningeal disease.
* Subject has had prior therapies with Dacarbazine (DTIC) or TMZ containing regimens.
* The subject has received an investigational agent within 28 days prior to study drug administration.
* Subject with a history of seizure disorder and currently receiving medications for seizure disorders (e.g., steroid or anticonvulsant drugs).
* The subject has had another active malignancy within the past 1 year with the exception of definitely treated carcinomas in situ, superficial bladder cancer, and non-melanoma carcinoma of the skin. Questions regarding inclusion of individual subjects should be discussed with the Abbott Medical Monitor.
* Clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * active uncontrolled infection,
  * symptomatic congestive heart failure,
  * unstable angina pectoris or cardiac arrhythmia,
  * Psychiatric illness/social situation that would limit compliance with study requirements,
  * Or any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities.
* Subject has previously been treated with a PARP inhibitor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Protein-specific antigen (PSA) test | Day 0 through investigator-determined discontinuation (final visit)
  This is performed to assess if ABT-888 combined with temozolomide has activity in patients with prostate cancer as reflected by the prostate-specific antigen (PSA).

SECONDARY OUTCOMES:
Assessment of Efficacy | Day 0 through investigator-determined discontinuation
  Evaluate the safety and tolerability of the combination therapy through safety assessments (i.e. electrocardiogram (ECG), clinical laboratory tests, vital signs, Adverse Event assessments, serious adverse events, physical exams, computed tomography (CT) scans)
Assessment of Safety | Day 0 through survival follow-up
  Assess the objective response rate (ORR), PSA decline, time to progression (TTP), progression free survival (PFS), and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Bhardwaj Desai, MD, Study Director — AbbVie

REFERENCES:
- [Result] Hussain M, Carducci MA, Slovin S, Cetnar J, Qian J, McKeegan EM, Refici-Buhr M, Chyla B, Shepherd SP, Giranda VL, Alumkal JJ. Targeting DNA repair with combination veliparib (ABT-888) and temozolomide in patients with metastatic castration-resistant prostate cancer. Invest New Drugs. 2014 Oct;32(5):904-12. doi: 10.1007/s10637-014-0099-0. Epub 2014 Apr 26. PMID 24764124